CLINICAL TRIAL: NCT03082885
Title: A Randomized Controlled Trial to Evaluate Efficacy and Safety of Thymosin-α1 Administration in Patients With HBV-related Acute-on-chronic Liver Failure
Brief Title: The Efficacy and Safety of Thymosin-α1 in Patients With HBV-related ACLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thymosin-α1
Record Dates: First submitted 2017-02-23; First posted 2017-03-17 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymosin-α1 group (Experimental): Patients receive treatment based on standard Therapy with additional Thymosin-α1
  Interventions: Drug: Thymosin-α1
- control group (No Intervention): Patients receive treatment based on standard Therapy

INTERVENTIONS:
Drug: Thymosin-α1 — 1.6 mg s.c injection once per day for 7 days, then 1.6 mg s.c injection twice a week for 11 weeks.
  Other Names: Zadaxin
  Arms: Thymosin-α1 group

SUMMARY:
A randomized controlled trial to evaluate efficacy and safety of Thymosin-α1 administration in patients with HBV-related Acute-on-chronic liver failure.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV)-related acute-on-chronic liver failure (ACLF) is a severe disease with high mortality. In this study, the investigators intend to assess the efficacy and safety of Thymosin-α1 in patients with HBV-related Acute-on-chronic liver failure.

ELIGIBILITY:
Inclusion Criteria:

* 1.Chronic hepatitis B.(Hepatitis B surface antigen positive for more than 6 months or having evidence of chronic hepatitis B virus infection).
* 2.Defined by an acute deterioration in transaminase greater than or equal to 5 times upper normal limit over14 days.
* 3.Development of jaundice (serum bilirubin greater than or equal to 10mg/dl).
* 4.Development of coagulopathy(PTA≤40% or INR≥1.5 ).
* More than one of the 5-8 criteria：
* 5.Development of hepatic encephalopathy.
* 6.Development of hepatorenal syndrome.
* 7.Hepatic narrowing progressively.
* 8.Development of massive ascites or peritonitis.
* 9. Willing to provide informed consent and comply with the test requirements

Exclusion Criteria:

* 1.Patients who have hepatocellular carcinoma confirmed by ultrasound/CT/MR.
* 2.Patients who have autoimmune disease (such as inflammatory bowel disease, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, etc ) or with abnormal elevation level of autoimmune antibody.
* 3.Model for end-stage liver disease (MELD) score <17 or >35.
* 4.Patients with significant co-morbid illnesses such as cardiovascular or respiratory or intrinsic renal diseases which by themselves may have a bearing on the outcome.
* 5.Patients with diseases that researchers consider inappropriate to participate in the study.
* 6.Patients who have disseminated intravascular coagulation.
* 7.Drug allergy.
* 8.Patients with any other contraindications to thymosin alpha1.
* 9.Patients who participated in other clinical trials at the same time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The liver transplantation-free survival rate of 90 days | 90 days
  Survival condition of the patients were observed for 90 days

SECONDARY OUTCOMES:
The liver transplantation-free survival rate of 180 days | 180 days
  Survival condition of the patients were observed for 180 days
Number of participants with ferver, bleeeding of injection site, amyotrophy and arthralgia | 24 weeks
  Fever, bleeeding of injection site, amyotrophy and arthralgia were observed during the treatment in both group.
Complications after 48 hours admission | 24 weeks
  Occurence of encephalopathy, infection, bleeding,hepatorenal syndrome after 48 hours admission.
Hepatitis B virus DNA load change | 24 weeks
  Hepatitis B virus DNA were measured on week 0, 4,8,12 and 24 after the start of the infusion in both groups
Causes of death/liver transplantation | 24 weeks
  Causes of death/liver transplantation (e.g. liver failure, multiple organs failure, severe infection) were recorded in both groups.
Inflammatory indexes change | 24 weeks
  Inflammatory indexes were measured on week0,1,2, 4,8,12 and 24 after the start of the infusion in both groups
Alanine aminotransferase change | 24 weeks
  Levels of alanine aminotransferase were measured on week0,1,2, 4,8, 12 and 24 after the start of the infusion in both groups
Glutamic oxaloacetic transaminase change | 24 weeks
  Levels of glutamic oxaloacetic transaminase were measured on week0,1,2, 4,8, 12 and 24 after the start of the infusion in both groups
Total bilirubin change | 24 weeks
  Levels of total bilirubin were measured on week0,1,2, 4,8,12 and 24 after the start of the infusion in both groups
Plasma thrombin time change | 24 weeks
  Levels of plasma thrombin time were measured on week0,1,2, 4,8,12 and 24 after the start of the infusion in both groups
Albumin time change | 24 weeks
  Levels of albumin were measured on week0,1,2, 4,8, 12 and 24 after the start of the infusion in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Lin B Liang, MD, Principal Investigator — leading
Locations (1):
- Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No